CLINICAL TRIAL: NCT04574791
Title: Addition of Muscle Relaxants in a Multimodal Analgesic Regimen for Analgesia After Primary Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAUS20d635
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — tizanidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Pain Regimen (No Intervention): current standard of care post-operative pain regimen in the hospital, which comprises of standing doses of oral acetaminophen 975 mg three times a day, gabapentin 300 mg two times a day, and intravenous ketorolac 30 mg three times a day for patients <65 years and 15 mg IV Q8h for patients who are >65 years, supplemented with PRN oxycodone and tramadol.
- Multimodal Pain Regimen + Tizanidine (Experimental): current standard of care post-operative pain regimen in the hospital, which comprises of standing doses of oral acetaminophen 975 mg three times a day, gabapentin 300 mg two times a day, and intravenous ketorolac 30 mg three times a day for patients <65 years and 15 mg IV Q8h for patients who are >65 years, supplemented with PRN oxycodone and tramadol supplemented with standing doses of oral tizanidine in the hospital and for 14 days after discharge
  Interventions: Drug: TiZANidine 2 MG Oral Capsule

INTERVENTIONS:
Drug: TiZANidine 2 MG Oral Capsule — Tizanidine 2 mg q8h (standing; # 42 tablets) + Multimodal pain regimen
  Arms: Multimodal Pain Regimen + Tizanidine

SUMMARY:
This is a prospective, cluster-randomized, two-arm, comparative study aimed at determining whether addition of tizanidine ( an oral muscle relaxant) to a multimodal pain regimen following primary TKA reduces opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* - Patients undergoing unilateral primary TKA with underlying diagnosis of osteoarthritis.
* ASA I - III
* Spinal anesthesia
* All patients will have a total knee arthroplasty utilizing a medial parapatellar approach with cruciate sacrificing implants and patellar resurfacing. A tourniquet will be used in all cases.
* Men and women between 18 and 80 years who are willing and able to provide informed consent

Exclusion Criteria:

* Opioid use greater than 10 mg/day morphine equivalents continuously for one month within 3 months preoperatively
* Inability to take/allergy to the protocol medications
* Contraindication to regional anesthesia
* Non-English speaking
* ASA IV or greater
* Psychiatric or cognitive disorders
* Allergy/contraindications to protocol medications.
* Renal insufficiency with Cr > 2.0 or hepatic failure
* Sensory/motor disorder involving the operative limb
* PCS score >20
* Patients with severe cardiac or neurological conditions precluding the use of study medications
* Patients using anticoagulation other than aspirin for the 14-day period after discharge

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
opioid consumption (MME) postoperatively | the first 14-days postoperatively
  Primary outcome is patients total opioid consumption for the first 14 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States